CLINICAL TRIAL: NCT05113160
Title: Understanding the Mechanisms of Change and Optimal Parameters in Conversation Treatment for Aphasia
Brief Title: Conversation Group Treatment for Aphasia: Does it Work?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Temple University (Other); Adler Aphasia Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4341E
Record Dates: First submitted 2021-09-29; First posted 2021-11-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Aphasia, Acquired
Keywords: aphasia; treatment; functional; communication; conversation group treatment; aphasia group; conversation treatment; communication disorder
MeSH Terms: conditions — Aphasia; Communication; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Parallel groups with delayed treatment control group.
Who Masked: Outcomes Assessor
Masking Description: Data coders will be blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment efficacy: Delayed Control Group (No Intervention): Treatment cycle 1 only.
- Experimental: Group Size x Aphasia Severity (Experimental): Outcomes will be measured for individuals who participate in large group (6-8 group members) compared to dyads (2 group members), and whether this relationship differs as a function of aphasia severity (severe vs. mild-moderate aphasia).
  Interventions: Behavioral: Conversation Treatment for Aphasia
- Experimental: Group composition (Experimental): Outcomes will be measured for individuals who participate in homogeneous compared to heterogeneous groups (6-8 people with aphasia), based on aphasia severity (severe vs. mild-moderate aphasia).
  Interventions: Behavioral: Conversation Treatment for Aphasia

INTERVENTIONS:
Behavioral: Conversation Treatment for Aphasia — Conversation treatment is a theoretically motivated approach in which a speech language pathologist facilitates discourse about topics of interest to the client using individualized, multi-modal supports. Treatment occurs either in groups of 6-8 people with aphasia or 2 people with aphasia. Individual communication goals are targeted for each group member within the context of naturalistic conversations.
  Arms: Experimental: Group Size x Aphasia Severity; Experimental: Group composition

SUMMARY:
The proposed research will test the efficacy of group conversation treatment for people with aphasia and explore whether the effects of treatment differ as a result of the following factors:

1. Group size: Do large groups of 6-8 people with aphasia or dyads of 2 people with aphasia demonstrate different levels of improvement with this treatment?
2. Group composition: Do effects of conversation group treatment differ if the groups include members with similar or different types of aphasia?
3. Aphasia severity: Do effects of conversation group treatment differ if the individuals within the group have mild-moderate or moderate-severe profiles of aphasia?

Treatment sessions will occur in groups of 6-8 people with aphasia or with 2 people with aphasia. During treatment sessions, discourse will be facilitated on a focused set of every day topics, such as current events or travel. Linguistic and multi modal cueing hierarchies will be tailored to individual client goals and used to maximize communication success.

The prediction is that conversation treatment is an effective method for improving communication in people with aphasia, but that specific benefits may differ based on variables such as group size, group composition, and aphasia severity. The results will help inform best practices for aphasia treatment and refine a hypothesized model about the mechanisms underlying conversation treatment.

DETAILED DESCRIPTION:
Aphasia is a language disorder that affects approximately two million Americans. The communication barriers associated with aphasia limit the ability to return to work and hobbies, worsen social relationships, and lead to social isolation. Social isolation is correlated with many negative health outcomes, including mortality. As a result, the consequences of aphasia can be wide reaching and severe. Group treatment has the potential to improve communication and reduce social isolation, while also reducing medical costs. However, this treatment format lacks a strong evidence base.

This research uses a hypothesis-driven approach to test the efficacy of conversation treatment and develop and refine a mechanistic pathway of how conversation treatment leads to behavioral changes in communication ability. We will systematically explore whether the effects of treatment differ as a result of number of participants (large group or dyad), group composition (heterogenous versus homogenous profiles of aphasia), and severity of aphasia. The study will enroll a total of 168 participants with aphasia across three sites. In cycle one, 72 participants will be randomly assigned to one of three conditions: dyad treatment, traditional group treatment or delayed control group. In cycles two and three, 48 participants with severe aphasia and 48 participants with mild-moderate aphasia will be randomly assigned to either large group or dyad conditions. In all cycles, treatment will occur for 60 minutes, twice per week for 10 weeks.

During treatment sessions, a speech pathologist will facilitate discourse on a focused set of salient topics, such as current events, using individualized, linguistic and multimodal cueing hierarchies. The primary outcome measure is a functional measure of communication (Aphasia Communication Outcome Measure, ACOM; Hula et al., 2015). Secondary outcome measures will include standardized tests and patient reported outcome measures, and examine linguistic and functional communication abilities. All participants will be assessed pre-, post-, 4 weeks post- and 12 weeks post-treatment.

The proposed research will address the following specific aims. Specific Aim 1 is to examine efficacy of conversation treatment delivered in dyads and large groups compared to a delayed-treatment control group. Specific Aim 2 is to determine optimal parameters for conversation treatment by testing whether the treatment effects differ as a function of aphasia severity (2A) or group composition (2B). Specific Aim 3 will test a hypothesized model of the pathway by which conversation treatment effects behavioral change. The results will provide further efficacy for conversation treatment and inform about the optimal parameters and outcomes of this intervention. This work takes a vital first step towards elucidating the mechanisms of change in conversation group treatment, with a long-term goal of ensuring access to cost-effective care for people with aphasia.

ELIGIBILITY:
Criteria for All Treatment Cycles:

Inclusion Criteria:

* Clinical diagnosis of aphasia
* At least 6 months post-onset of stroke in the language-dominant hemisphere.
* Native English speakers
* Demonstrate sufficient auditory comprehension skills to participate in a supported conversation, based on results of standardized aphasia tests

Exclusion

* No history of neurological disease (other than stroke)
* No history of developmental speech, language, or learning disabilities
* No current serious medical illness (e.g., cancer)
* Participants will be asked to abstain from concurrent speech language treatment.

Separate criteria for Treatment Cycles 1, 2, and 3 based on aphasia severity:

Cycle 1 Severity-based Inclusion Criteria (Completed 2022):

-- All aphasia profiles and severity levels.

Cycle 2 Severity-based Inclusion Criteria (Completed 2023):

-- Participants with severe aphasia

Cycle 3 Severity-based Inclusion Criteria (Completed 2024):

-- Participants with mild-moderate aphasia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Scores on Aphasia Communication Outcome Measure from Pre- to Post- Treatment | Baseline and up to 12 weeks after baseline
  The Aphasia Communication Outcome Measure (ACOM; Hula et al, 2015) is a patient reported outcome measure that reflects the clinical endpoint of conversation treatment. The ACOM is a psychometrically validated measure of the impact of aphasia on communication in daily life. The ACOM asks questions such as how effectively the person with aphasia talks to family members or clerks in a store. Standardized scores (T-scores) are computed, with higher values indicating better self-reported communication ability.
Change in Scores on Aphasia Communication Outcome Measure from Pre-Treatment to One month Post-Treatment | Baseline and up to 16 weeks after baseline
  The Aphasia Communication Outcome Measure (ACOM; Hula et al, 2015) is a patient reported outcome measure that reflects the clinical endpoint of conversation treatment. The ACOM is a psychometrically validated measure of the impact of aphasia on communication in daily life. The ACOM asks questions such as how effectively the person with aphasia talks to family members or clerks in a store. Standardized scores (T-scores) are computed, with higher values reflecting better self-reported communication ability.

SECONDARY OUTCOMES:
Change in Scores on Comprehensive Aphasia Test from Pre- to Post- Treatment | Baseline and up to 12 weeks after baseline
  The Comprehensive Aphasia Test (CAT; Swinburn, Howard, & Porter, 2004) is a standardized test battery that targets expressive and receptive language in the oral and written modalities. Six sections of the language battery will be administered: comprehension of spoken language, comprehension of written language, repetition, naming, oral reading, and spoken picture description. Standardized scores (T-scores) are computed, with higher values reflecting better outcomes.
Change in Scores on Comprehensive Aphasia Test from Pre-Treatment to One month Post-Treatment | Baseline and up to 16 weeks after baseline
  The Comprehensive Aphasia Test (CAT; Swinburn, Howard, & Porter, 2004) is a standardized test battery that targets expressive and receptive language in the oral and written modalities. Six sections of the language battery will be administered: comprehension of spoken language, comprehension of written language, repetition, naming, oral reading, and spoken picture description. Standardized scores (T-scores) are computed, with higher values reflecting better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hoover, PhD, Principal Investigator — Boston University; Gayle DeDe, PhD, Principal Investigator — Temple University
Locations (3):
- United States (3):
  - Boston University - Charles River Campus, Boston, Massachusetts
  - Adler Aphasia Center, Maywood, New Jersey
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT05113160/ICF_002.pdf